CLINICAL TRIAL: NCT03633487
Title: A Phase I, Open-label, Single-dose, Single Period Study to Evaluate the Pharmacokinetics of Mucinex® 1200 mg Extended-Release Bi-layer Tablet in Normal Healthy Subjects.
Brief Title: Study to Evaluate the Pharmacokinetics of Mucinex® 1200 mg Extended-Release Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-MUC-05
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Acetylcysteine; Guaifenesin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mucinex® 1200 mg (Experimental): Mucinex® 1200 mg Extended-Release (ER) Bi-Layer tablet (single dose)
  Interventions: Drug: Mucinex®

INTERVENTIONS:
Drug: Mucinex® — Mucinex® 1200 mg ER Bi-Layer tablet
  Other Names: guaifenesin

SUMMARY:
Characterize and assess PK of guaifenesin in Mucinex® 1200 mg ER Bi-Layer Tablet

DETAILED DESCRIPTION:
A Phase I, Open-Label, Single-Dose, Single Period Study to Evaluate the Pharmacokinetics of Mucinex® 1200 mg Extended-Release Bi-Layer Tablet in Normal Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥19 to 55 years of age inclusive.

   All females who were of childbearing potential must have been using one of the following acceptable birth control methods for the time periods specified:
   1. Intrauterine device (IUD) in place for at least 3 months prior to Day 1 through 30 days beyond study completion.
   2. Barrier method (condom or diaphragm) with spermicide for at least 7 days prior to screening through 30 days beyond study completion.
   3. Stable hormonal contraceptive (oral, depo injection, transdermal patch, or vaginal ring) for at least 3 months prior to Day 1 through 30 days beyond completion of study.

   Note: Abstinence (sexually inactive) was not an acceptable form of contraception; however, abstinent female subjects could have been admitted to the study if they had reported being abstinent at least 14 days prior to screening and they agreed, and signed an "Abstinence Statement" to the effect, that upon becoming sexually active, they would use a condom with spermicide from that time through 30 days beyond completion of the study.

   Females of non-childbearing potential must have been surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to Day 1 or hysterectomy and/or bilateral oophorectomy at least 3 months prior to Day 1 or post-menopausal ≥2 years prior to Day 1). A follicle stimulating hormone level (FSH) >40 mIU/mL must have been obtained and in the record for any post-menopausal female.
2. Negative serum pregnancy test at Screening and at Check-in for all female subjects.
3. Good general health as determined by the PI's review of medical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements (after 2 minutes resting in the seated position), and clinical laboratory measures.
4. Body mass index (BMI) of 19 to 29 kg/m2, inclusive. (BMI = weight (kg)/[height (m2)]).
5. Non-tobacco users, who had not used nicotine or nicotine-containing products for at least 6 months prior to Day 1.
6. Negative finding on tests for Hepatitis B surface antigen (HBsAG), Hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV).
7. Negative urine screen for drugs of abuse and alcohol at Screening and at Check-in.
8. Likely to be compliant with study requirements and complete the study, as determined by the Investigator.
9. Able to read, understand, and sign the informed consent after the nature of the study had been explained and had read, signed, and dated an Institutional Review Board (IRB)-approved informed consent form for subjects to participate in the study.

Exclusion Criteria:

1. Clinically significant abnormalities detected by medical history, physical examination, vital sign measurements, ECG findings, or clinical laboratory findings (as determined by the PI). If the subject's hemoglobin dropped below 11.0 gm/dL during the study, the subject may have been dropped from the study at the discretion of the PI/designee.
2. Any disease or condition, which could impact absorption, distribution, metabolism, or elimination of the study drug (as determined by the PI/designee).
3. Females who were pregnant or nursing.
4. History of hypersensitivity reaction to guaifenesin.
5. Receipt of an investigational drug within 30 days prior to Day 1.
6. Abnormal diet (for whatever reason) during the 30 days prior to Day 1.
7. Donation of blood or significant loss of blood within 56 days prior to Day 1.
8. Donation of plasma within 14 days prior to Day 1.
9. Known or suspected use of illicit drugs (i.e., opiates, barbiturates, marijuana, et. al.).
10. The use of any medication, prescription or over-the-counter (OTC) (including herbal supplements) within the 14 days or 5 half-lives of the drug (whichever was longer) prior to Day 1 (with the exception of hormonal contraceptives for women of child-bearing potential).
11. Alcoholism or medicinal product or drug abuse within the past two years or excessive alcohol consumption (more than 10 units per week) [one unit is defined as 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of spirits (i.e., "hard" liquor such as gin, whiskey, or vodka, et. al.)]. The subject was not to experience tolerance, withdrawal, compulsive use, or substance related problems such as medical complications, disruption in social and family relationships, vocational or financial difficulties, or legal problems.
12. Consumption of grapefruit, pummelo, Seville orange, or grapefruit juice within 14 days prior to dosing on Day 1 through study completion.
13. Consumption of alcohol within the 48 hours prior to dosing on Day 1.
14. Persons involved directly with the conduct of this study (i.e., Investigator, Sub-Investigators, Study Coordinators, etc.) or employees of Reckitt Benckiser and their families.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2011-10-15 (Actual); Study Completion 2011-10-15 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study.
Pre-assignment Details: A total of 24 subjects entered the study; All 24 subjects were included single-period.
Groups:
- Mucinex® 1200 mg: Single dose Mucinex® 1200 mg Extended-Release (ER) Bi-Layer tablet by mouth.
Period: Overall Study
Arm/Group | Mucinex® 1200 mg
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Race [Number; unit: participants]
  Asian | 1
  Black or African American | 1
  White | 22
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
Weight [Mean (Standard Deviation); unit: kg] | 75.42 (12.711)
Height [Mean (Standard Deviation); unit: cm] | 175.8 (9.65)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 24.220 (2.4480)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Pharmacokinetic Parameters (Cmax) Maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 1,2,3,4,5,6,7, 8, 9, 10, 11, 12, 13, 14, 15, 20, 25, 30, 35, 40, 45, 50, and 55 minutes; 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 5, 6, 7, 8, 10, 12, 14, 16 and 24 hours on Day 1
Population: Pharmacokinetic (PK) population includes subjects with at least one PK sample. Available data from any subjects who vomited within 12 hours after dosing were to be included in the PK data sets.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 24
ng/mL | 1634 (769.95)

2. Primary Outcome: Time of the Maximum Observed Plasma Concentration (Tmax)
Description: Pharmacokinetic Parameter (Tmax) Time of the maximum observed plasma concentration
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 24
hr | 0.9753 (0.61407)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-t)
Description: Pharmacokinetic Parameter (AUC0-t) is Area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 24
ng*hr/mL | 6515.5 (2765.33)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf)
Description: Pharmacokinetic Parameter (AUC0-inf) Area under the plasma concentration versus time curve from time 0 to infinity.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 23
ng*hr/mL | 6733.5 (2831.57)

5. Primary Outcome: Percentage of AUC0-inf Extrapolated Area Under Plasma Concentration Curve Ratio (AUCR) of Guaifenesin
Description: Pharmacokinetic Parameter (AUC%extrap) Percent of AUC0-inf extrapolated AUCR = 100 - (AUC0-t/ AUC0-inf) x 100
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of AUC0-inf extrapolated AUCR
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 23
Percentage of AUC0-inf extrapolated AUCR | 1.950 (2.7458)

6. Primary Outcome: Apparent First-order Terminal Elimination Rate Constant (Kel)
Description: Pharmacokinetic Parameter (Kel) Apparent first-order terminal elimination rate constant
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 23
1/hr | 0.2644 (0.16374)

7. Primary Outcome: Terminal Elimination Half Life (t1/2)
Description: Pharmacokinetic Parameter (t1/2) is Apparent terminal elimination half-life.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 23
hr | 3.374 (1.6383)

8. Primary Outcome: Time at Which the Percentage of Subjects Achieved a Target Concentration of at Least 65 ng/mL (T65)
Description: Pharmacokinetic Parameter (T65) is te time when guaifenesin plasma concentration achieved a target concentration of at least 65 ng/mL.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 24
hr | 0.1999 (0.10427)

9. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs)
Description: Intensity was determined by the Investigator. For symptomatic adverse events (AEs) the following definitions were applied.
  Mild = AE did not limit usual activities; subject may have experienced slight discomfort.
  Moderate = AE resulted in some limitation of usual activities; subject may have experienced significant discomfort.
  Severe = AE resulted in an inability to carry out usual activities; subject may have experienced intolerable discomfort/pain.
  Relationship to Investigational Medicinal Products (IMP) Unlikely = Slight, but remote, chance that AE was caused by IMP. Possible = Reasonable suspicion that the AE was caused by IMP. Probable = Most likely that AE was caused by IMP.
Time Frame: Up to Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mucinex® 1200 mg
Number analyzed (Participants) | 24
Participants
  TEAE by severity: Mild | 3
  TEAE by severity: Moderate | 0
  TEAE by severity: Severe | 0
  Relationship to IMP - Definite | 0
  Relationship to IMP - Probable | 0
  Relationship to IMP - Possible | 1
  Relationship to IMP - Unlikely | 0
  Relationship to IMP - None | 2

ADVERSE EVENTS:
Time Frame: Up to Day 2
Arm/Group | Mucinex® 1200 mg
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mucinex® 1200 mg (N=24)
Catheter site swelling (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No